CLINICAL TRIAL: NCT01209871
Title: Phase I Study of an Active Immunotherapy for Asymptomatic Phase Lymphoplasmacytic Lymphoma With DNA Vaccines Encoding Antigen-Chemokine Fusion
Brief Title: Vaccine Therapy in Treating Patients With Lymphoplasmacytic Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0465; NCI-2012-01897 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2010-02091 (Other: CTRP (Clinical Trial Reporting Program)); 2009-0465 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Lymphoplasmacytic Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (vaccine therapy) (Experimental): Patients receive autologous lymphoma immunoglobulin-derived scFV-chemokine DNA vaccine ID at 0, 4, and 8 weeks.
  Interventions: Biological: Autologous Lymphoma Immunoglobulin-derived scFv-chemokine DNA Vaccine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Autologous Lymphoma Immunoglobulin-derived scFv-chemokine DNA Vaccine — Given ID
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of vaccine therapy in treating patients with lymphoplasmacytic lymphoma. Vaccines made from a person's cancer cells may help the body build an effective immune response to kill cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and feasibility of using a novel lymphoma deoxyribonucleic acid (DNA) vaccine encoding macrophage inflammatory protein 3 alpha (MIP3a)-fused lymphoma idiotype in single chain format.

II. To determine the maximum tolerated dose (MTD) of the vaccine.

SECONDARY OBJECTIVES:

I. To assess the immunogenicity of the vaccine to generate tumor-specific cellular and humoral immune responses.

OUTLINE: This is a dose-escalation study.

Patients receive autologous lymphoma immunoglobulin-derived single-chain variable fragment (scFV)-chemokine DNA vaccine intradermally (ID) at 0, 4, and 8 weeks.

After completion of study treatment, patients are followed up at 4 weeks, and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Tissue diagnosis of lymphoplasmacytic lymphoma with surface immunoglobulin G (IgG), immunoglobulin A (IgA) or immunoglobulin M (IgM) phenotype with a monoclonal heavy and light chain as determined by flow cytometry; all primary diagnostic lymph node and/or bone marrow biopsies will be reviewed at the University of Texas M.D. Anderson Cancer Center (UTMDACC)
* Previously untreated patients with lymphoplasmacytic lymphoma (of any subtype: IgG, IgA, IgM) in the asymptomatic phase
* Patients must provide a lymph node sample of at least 1.5 cm in the long axis, or a bone marrow aspiration sample providing at least 5 million cluster of differentiation (CD)20 and/or CD38+ (approximately 10 ml)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Serum creatinine =< 1.5 mg/dl and a creatinine clearance >= 30 ml/min
* Total bilirubin =< 1.5 mg/dl unless felt secondary to Gilbert's disease
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2 x upper limit of normal
* Ability to provide informed consent, and to return to clinic for adequate follow-up for the period that the protocol requires
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study and for 30 days after the last vaccination has been administered
* Male subject agrees to use an acceptable method for contraception for the duration of the study

Exclusion Criteria:

* Human immunodeficiency virus (HIV), hepatitis B and/or hepatitis C infection
* Pregnancy or lactating females
* Patients with previous history of malignancy within the last 5 years except curatively treated squamous or basal cell carcinoma of the skin or curatively treated carcinoma in-situ of other organs
* Any medical or psychiatric condition that in the opinion of the principal investigator would compromise the patient's ability to tolerate this treatment
* Patients with New York Heart Association class 3 or 4 disease
* Patients with a history of autoimmune diseases except for Hashimoto's thyroiditis
* Patients with positive antinuclear antibody (ANA) and/or anti-double strand (ds) DNA antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-02-26 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose defined as the highest dose level in which 6 patients have been treated with less than 2 instances of dose limiting toxicity according to the National Cancer Institute Common Toxicity Criteria version 4.0 | 4 weeks
  Toxicity type and severity will be summarized by frequency tables.

SECONDARY OUTCOMES:
Immune response defined as at least a three-fold rise in the precursor frequency of tumor-reactive T cells | At 12 weeks
  The rate of immune response will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Sheeba Thomas, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Thomas SK, Cha SC, Smith DL, Kim KH, Parshottam SR, Rao S, Popescu M, Lee VY, Neelapu SS, Kwak LW. Phase I study of an active immunotherapy for asymptomatic phase Lymphoplasmacytic lymphoma with DNA vaccines encoding antigen-chemokine fusion: study protocol. BMC Cancer. 2018 Feb 13;18(1):187. doi: 10.1186/s12885-018-4094-2. PMID 29439670
- See also: MD Anderson Cancer Center — http://www.mdanderson.org